CLINICAL TRIAL: NCT00651625
Title: Randomized Controlled Trial of the Reciprocating Procedure Device Versus the Conventional Syringe in Syringe-and-Needle Procedures
Brief Title: Reciprocating Medical Devices - a Study of a New Safety Device
Acronym: RPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRRC 04-347; HRRC 04-347 (Other Grant/Funding Number: University of New Mexico); 04-347 (Other: University of New Mexico)
Record Dates: First submitted 2008-03-21; First posted 2008-04-03 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Trauma; Thyroid Nodule; Cancer
Keywords: arthrocentesis; injections; anesthesia; biopsy; aspiration; syringe; safety; pain
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Wounds and Injuries; Thyroid Nodule; Neoplasms; Pain | interventions — Syringes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The intervention is the use of the reciprocating procedure device (RPD) (AVANCA Re No. 1091001) (intervention) (Arm 1) with and without ultrasound guidance (intervention) in a syringe and needle procedure in comparison to a conventional syringe (BD Ref 309604) (control, Arm 2).
  Interventions: Device: Reciprocating Procedure Device (RPD) - AVANCA Re No. 1091001
- 2 (Active Comparator): The conventional syringe (BD Ref 309604) is used to performed the syringe and needle procedure and outcome (effect of procedure (pain scores at 2 weeks and 6 months compared to preprocedural pain scores), and procedural pain (pain scores during procedure) are determined) and compared to Arm 1.
  Interventions: Device: conventional syringe - BD Ref 309604

INTERVENTIONS:
Device: Reciprocating Procedure Device (RPD) - AVANCA Re No. 1091001 — The RPD is a safety syringe device that is hypothesized to be safer, less painful, and more effective for patients undergoing a syringe and needle procedure (please see arm #1).
  Other Names: AVANCA RPD
  Arms: 1
Device: conventional syringe - BD Ref 309604 — the conventional syringe or the RPD will be used for syringe and needle procedures performed by physicians.
  Other Names: syringe; conventional syringe; traditional syringe
  Arms: 2

SUMMARY:
The study design is a randomized study to directly compare the performance and the outcome of syringe and needle procedures with a standard syringe or the new reciprocating procedure device (RDP), which is a type of safety syringe. Over a 5 year period, 820 subjects who require and assent to a syringe and needle procedure for their usual and customary care will be randomized to either a conventional syringe or the RPD with one arm with and without ultrasound guidance. The RPD is designed to be safer, faster, less painful, and more effective for the patient, and the mechanics of the RPD are intended to provide the physician with better needle control, resulting in less needle trauma to patient tissues, and thus, reduced bleeding and pain for the patient. This clinical trial will address whether the RPD is indeed superior to the conventional syringe for shots, injections, and needle procedures, and whether it is a safer, less painful syringe.

DETAILED DESCRIPTION:
* BACKGROUND

The syringe is an ancient device designed principally to inject medications. However, because of the inherent biomechanics of the human hand and the interaction of the hand with the piston, the syringe is very stable and easily controlled the injection phase, but is extremely unstable and difficult to control in the aspiration phase. New reciprocating technology that accommodates the biomechanics of hand function has great promise of improving the stability and safety of hand-held devices, including procedure syringes.

* EXPERIMENTAL DESIGN AND METHODS

The study design is a randomized study to directly compare the performance and the outcome of syringe and needle procedures accomplished either with a standard syringe or the new reciprocating procedure device (RDP). Over a 5 year period, 820 subjects who require and assent to a syringe procedure for their usual and customary care will be randomized to either a conventional syringe or the reciprocating syringe. The following syringe procedures will be studied: 1) local anesthesia, 2) centesis (arthrocentesis, paracentesis, thoracentesis, amniocentesis, pericardiocentesis), 3) aspiration and puncture (aspiration of bursa, cyst, abscess, shunt, bone marrow, and other syringe aspiration procedures), 4) injection of a therapeutic or diagnostic substance into a joint, bursa, vessel, or other body structure, 5) fine needle biopsy with syringe vacuum of a mass or tissue, 6) irrigation procedures (wound, bladder, and other irrigation procedures), and 7) vascular access (introduction of a wire, catheter, or sheath into a blood vessel), and 8) with and without ultrasound guidance.

In a subject with multiple individual procedure sites, or requires multiple separate biopsies, each will be randomized between the two syringes, and each biopsy or fluid sample will be analyzed separately (as is medically appropriate). The physicians who will perform the syringe procedures will be those physicians who usually perform the syringe procedures and are credentialed to do so. Outcome data collection will occur first by one of the investigators observing the procedure and collecting the data by real time interview and by chart review including cost analysis. Outcome data will include effectiveness (preprocedural pain, pain at 2 weeks post procedure, and pain at 6 months postprocedure), procedure time, patient pain, operator satisfaction, trauma to tissues, complications, diagnostic yield, overall medical care costs and hospital stay. Retrospective review of 30 charts of the device used clinically has also been approved (2006). Analysis of data will be performed by a statistician blinded to treatment group.

*SIGNIFICANCE: The proposed study will be the first to study the clinical performance characteristics of a medical device that incorporates the new reciprocating technology designed to take advantage of the inherent biomechanical stability characteristics of the human hand. The preclinical studies presented in the preliminary data demonstrate markedly enhanced device performance characteristics, and much greater control and stability, strongly suggesting that reciprocating devices will be safer, more effective, more economical, and provide better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A syringe and needle procedure is required for the normal customary care of the patient

Exclusion Criteria:

* hemorrhagic diathesis,
* use of anticoagulants and antiplatelet agents child or susceptible population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2004-11; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilmer L Sibbitt, Jr., MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sibbitt RR, Palmer DJ, Sibbitt WL Jr. Reciprocating procedure device for thyroid cyst aspiration and ablative sclerotherapy. J Laryngol Otol. 2009 Mar;123(3):343-5. doi: 10.1017/S0022215108003551. Epub 2008 Sep 17. PMID 18796180
- [Background] Sibbitt RR, Sibbitt WL Jr, Palmer DJ, Bankhurst AD. Needle aspiration of peritonsillar abscess with the new safety technology: the reciprocating procedure device. Otolaryngol Head Neck Surg. 2008 Aug;139(2):307-9. doi: 10.1016/j.otohns.2008.04.003. No abstract available. PMID 18656735
- [Background] Sibbitt RR, Palmer DJ, Sibbitt WL Jr. Integration of patient safety technologies into sclerotherapy for varicose veins. Vasc Endovascular Surg. 2008 Oct-Nov;42(5):446-55. doi: 10.1177/1538574408318479. Epub 2008 Jun 25. PMID 18583303
- [Background] Moorjani GR, Bedrick EJ, Michael AA, Peisajovich A, Sibbitt WL Jr, Bankhurst AD. Integration of safety technologies into rheumatology and orthopedics practices: a randomized, controlled trial. Arthritis Rheum. 2008 Jul;58(7):1907-14. doi: 10.1002/art.23499. PMID 18576358
- [Background] Sibbitt RR, Palmer DJ, Bankhurst AD, Sibbitt WL Jr. Integration of new safety technologies for needle aspiration of breast cysts. Arch Gynecol Obstet. 2009 Mar;279(3):285-92. doi: 10.1007/s00404-008-0710-8. Epub 2008 Jun 21. PMID 18568356
- [Background] Moorjani GR, Michael AA, Peisajovich A, Park KS, Sibbitt WL Jr, Bankhurst AD. Patient pain and tissue trauma during syringe procedures: a randomized controlled trial. J Rheumatol. 2008 Jun;35(6):1124-9. Epub 2008 Apr 15. PMID 18412301
- [Background] Sibbitt RR, Sibbitt WL Jr, Nunez SE, Kettwich LG, Kettwich SC, Bankhurst AD. Control and performance characteristics of eight different suction biopsy devices. J Vasc Interv Radiol. 2006 Oct;17(10):1657-69. doi: 10.1097/01.RVI.0000236837.47302.8E. PMID 17057008
- [Background] Gerstein NS, Martin HB, Toma, G MD; Sibbitt RR, Sibbitt WL Jr.. Central venous access with the new safety technology the reciprocating procedure device. Journal Clinical Anesthesiology 2008 (In Press).
- [Result] Bankhurst AD, Nunez SE, Draeger HT, Kettwich SC, Kettwich LG, Sibbitt WL Jr. A randomized controlled trial of the reciprocating procedure device for intraarticular injection of corticosteroid. J Rheumatol. 2007 Jan;34(1):187-92. PMID 17143968
- [Result] Nunez SE, Draeger HT, Rivero DP, Kettwich LG, Sibbitt WL Jr, Bankhurst AD. Reduced pain of intraarticular hyaluronate injection with the reciprocating procedure device. J Clin Rheumatol. 2007 Feb;13(1):16-9. doi: 10.1097/01.rhu.0000256280.85507.bd. PMID 17278943
- [Result] Nunez SE, Bedrick EJ, Kettwich SC, Kettwich LG, Bankhurst AD, Sibbitt WL Jr. A randomized, controlled trial of the reciprocating procedure device for local anesthesia. J Emerg Med. 2008 Aug;35(2):119-25. doi: 10.1016/j.jemermed.2007.08.060. Epub 2008 Feb 20. PMID 18281176
- [Result] Draeger HT, Twining JM, Johnson CR, Kettwich SC, Kettwich LG, Bankhurst AD. A randomised controlled trial of the reciprocating syringe in arthrocentesis. Ann Rheum Dis. 2006 Aug;65(8):1084-7. doi: 10.1136/ard.2005.045781. Epub 2005 Dec 8. PMID 16339287
- [Result] Sander O. Intra-articular corticosteroid injections with the reciprocating procedure device reduced procedural pain and duration more than the conventional syringe. Evid Based Med. 2007 Aug;12(4):106. doi: 10.1136/ebm.12.4.106. No abstract available. PMID 17885154
- [Result] Sibbitt W Jr, Sibbitt RR, Michael AA, Fu DI, Draeger HT, Twining JM, Bankhurst AD. Physician control of needle and syringe during aspiration-injection procedures with the new reciprocating syringe. J Rheumatol. 2006 Apr;33(4):771-8. Epub 2006 Mar 1. PMID 16511940
- [Result] Park KS, Peisajovich A, Michael AA, Sibbitt WL Jr, Bankhurst AD. Should local anesthesia be used for arthrocentesis and joint injections? Rheumatol Int. 2009 Apr;29(6):721-3. doi: 10.1007/s00296-008-0785-3. Epub 2008 Nov 27. No abstract available. PMID 19037606
- [Result] Michael AA, Moorjani GR, Peisajovich A, Park KS, Sibbitt WL Jr, Bankhurst AD. Syringe size: does it matter in physician-performed procedures? J Clin Rheumatol. 2009 Mar;15(2):56-60. doi: 10.1097/RHU.0b013e31819c1fc4. PMID 19265345
- [Derived] Kettwich LG, Sibbitt WL Jr, Emil NS, Ashraf U, Sanchez-Goettler L, Thariani Y, Bankhurst AD. New device technologies for subcutaneous fat biopsy. Amyloid. 2012 Jun;19(2):66-73. doi: 10.3109/13506129.2012.666508. Epub 2012 Mar 27. PMID 22452536
- [Derived] Sibbitt WL Jr, Michael AA, Poole JL, Chavez-Chiang NR, Delea SL, Bankhurst AD. Nerve blocks at the wrist for painful injections of the palm. J Clin Rheumatol. 2011 Jun;17(4):173-8. doi: 10.1097/RHU.0b013e31821bfed0. PMID 21617556
- [Derived] Hayward WA, Haseler LJ, Kettwich LG, Michael AA, Sibbitt Wl Jr, Bankhurst AD. Pressure generated by syringes: implications for hydrodissection and injection of dense connective tissue lesions. Scand J Rheumatol. 2011;40(5):379-82. doi: 10.3109/03009742.2011.560892. Epub 2011 Apr 6. PMID 21469942
- [Derived] Chavez-Chiang CE, Sibbitt WL Jr, Band PA, Chavez-Chiang NR, DeLea SL, Bankhurst AD. The highly accurate anteriolateral portal for injecting the knee. Sports Med Arthrosc Rehabil Ther Technol. 2011 Mar 30;3(1):6. doi: 10.1186/1758-2555-3-6. PMID 21447197
- [Derived] Ricciardi M, Roldan C, Sibbitt R, Sibbitt W Jr, Michael A, Palmer D. Highly controlled vascular syringes for pericardiocentesis. J Invasive Cardiol. 2010 Dec;22(12):580-4. PMID 21127362
- [Derived] Sibbitt WL Jr, Band PA, Chavez-Chiang NR, Delea SL, Norton HE, Bankhurst AD. A randomized controlled trial of the cost-effectiveness of ultrasound-guided intraarticular injection of inflammatory arthritis. J Rheumatol. 2011 Feb;38(2):252-63. doi: 10.3899/jrheum.100866. Epub 2010 Nov 15. PMID 21078710
- [Derived] Sibbitt RR, Palmer DJ, Sibbitt WL Jr, Bankhurst AD. Image-directed fine-needle aspiration biopsy of the thyroid with safety-engineered devices. Cardiovasc Intervent Radiol. 2011 Oct;34(5):1006-13. doi: 10.1007/s00270-010-0013-x. Epub 2010 Nov 6. PMID 21057794
- [Derived] Sibbitt WL Jr, Peisajovich A, Michael AA, Park KS, Sibbitt RR, Band PA, Bankhurst AD. Does sonographic needle guidance affect the clinical outcome of intraarticular injections? J Rheumatol. 2009 Sep;36(9):1892-902. doi: 10.3899/jrheum.090013. Epub 2009 Jul 31. PMID 19648304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: dates from 2004 to August 2010, recruited from medical clinic
Pre-assignment Details: patients recruited immediately at point of contact
Groups:
- 1Conventional Syringe: The intervention is the use of the reciprocating procedure device (RPD) with and without ultrasound guidance in a syringe and needle procedure in comparison to a conventional syringe. The RPD is used to performed the syringe and needle procedure and outcome (effect of procedure (pain scores at 2 weeks and 6 months compared to preprocedural pain scores), and procedural pain (pain scores during procedure) - are determined. Thus, pain scores as measured by the standard 10 cm Visual Analogue Pain Score are used to primary outcome as is standard in the field of pain. These scores from the two treatment arms are then compared statistically with each other by appropriate methods. It is hypothesized that the RPD will be more effective (reduced pain scores at 2 weeks and 6 months) and less pain (reduced procedural pain scores) compared to the same procedure with the conventional syringe.
- 2RPD Syring: Conventional Syringe - The conventional syringe is used to performed the syringe and needle procedure and outcome (effect of procedure (pain scores at 2 weeks and 6 months compared to preprocedural pain scores), and procedural pain (pain scores during procedure) are determined). The comparison is with the same procedure performed with the RPD syringe with and without ultrasound. It is hypothesized that the RPD will be more effective (reduced pain scores at 2 weeks and 6 months) and less pain (reduced procedural pain scores) compared to the same procedure with the conventional syringe.
Period: Overall Study
Arm/Group | 1Conventional Syringe | 2RPD Syring
Started | 219 | 218
Completed | 219 | 218
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1Conventional Syringe | 2RPD Syring | Total
Number analyzed (Participants) | 219 | 218 | 437
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 219 | 218 | 437
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (9.7) | 51.7 (14.8) | 52.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 177 | 352
  Male | 44 | 41 | 85
Region of Enrollment [Number; unit: participants]
  United States | 219 | 218 | 437

OUTCOME MEASURES:

1. Primary Outcome: Pain Using VAS (Visual Analogue Pain Scale)
Description: 0-10 cm VAS pain scale at 2 weeks compared to 0-10 cm VAS pain scale at 0 weeks where 0= no pain, and 10 = the worst pain imaginable. The difference (2 week VAS-0 week VAS) is the primary outcome measure.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cm
Groups:
- 2RPD Syringe: Conventional Syringe - The conventional syringe is used to performed the syringe and needle procedure and outcome (effect of procedure (pain scores at 2 weeks and 6 months compared to preprocedural pain scores), and procedural pain (pain scores during procedure) are determined). The comparison is with the same procedure performed with the RPD syringe with and without ultrasound. It is hypothesized that the RPD will be more effective (reduced pain scores at 2 weeks and 6 months) and less pain (reduced procedural pain scores) compared to the same procedure with the conventional syringe.
Arm/Group | 1Conventional Syringe | 2RPD Syringe
Number analyzed (Participants) | 219 | 218
cm | 5.2 (2.7) | 6.2 (2.9)

2. Secondary Outcome: Aspirated Fluid Volume
Description: Aspirated fluid volume during procedure
Time Frame: during procedure
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | 1Conventional Syringe | 2RPD Syringe
Number analyzed (Participants) | 219 | 218
ml | 7.2 (3.1) | 14.5 (4.1)

3. Secondary Outcome: Adverse Outcomes (Hemorrhage, Infection, Hematoma, Extravasation)
Time Frame: during procedure, 2 weeks afterwards, and 6 months afterwards
Measure: Number; unit: participants
Arm/Group | 1Conventional Syringe | 2RPD Syringe
Number analyzed (Participants) | 219 | 218
participants | 0 | 0

4. Secondary Outcome: Physician Satisfaction
Description: 0- 10 cm visual analogue satisfaction scale (VASS)
  0-10 cm VASS at 2 weeks compared to 0-10 cm VASS pain scale at 0 weeks where 0= completely dissatisfied, and 10 = completely satsified. The difference (2 week VAS-0 week VAS) is the outcome measure
Time Frame: during procedure
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 1Conventional Syringe | 2RPD Syringe
Number analyzed (Participants) | 219 | 218
cm | 6.4 (2.1) | 8.5 (3.1)
Statistical Analysis 1: Comparison: 1Conventional Syringe vs 2RPD Syringe; group comparisons using t-test and confidence intervals; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; non-applicable

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 1Conventional Syringe | 2RPD Syring
Serious Adverse Events (participants affected / at risk) | 0/219 | 0/218
Other Adverse Events (participants affected / at risk) | 0/219 | 0/218
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1Conventional Syringe (N=219) | 2RPD Syring (N=218)
(Investigations) | 0 (0) | 0 (0) — No adverse events

LIMITATIONS AND CAVEATS:
no adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No